CLINICAL TRIAL: NCT00394667
Title: Effect of Tesofensine on Weight Reduction in Patients With Obesity. A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Study.
Brief Title: Effect of Tesofensine on Weight Reduction in Patients With Obesity.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroSearch A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIPO-1
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tesofensine

INTERVENTIONS:
Drug: Tesofensine

SUMMARY:
Purpose:

To evaluate the efficacy on weight reduction, metabolic parameters and safety of tesofensine versus placebo in obese patients

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with 30 kg/m² ≤ BMI ≤ 40 kg/m²
* Males and females 18 to 65 years of age, extremes included
* Patients continuously receiving diet therapy as well as instructions on exercise at least for 2 weeks run-in, who during the run-in before randomization do not gain weight (< 2 kg)
* Females of childbearing potential must be non-pregnant and use safe contraceptive methods (the pill, IUD or surgically sterilized)
* Patients should be able to comply with study procedures
* Smoking habits should have been stable for at least 2 months
* Patients giving written informed consent

Exclusion Criteria:

* Use of prescription medication as listed
* Positive serum pregnancy test for women of childbearing potential
* Pregnant or lactating women, or women who are planning to become pregnant within the next 8 months
* Patients with specific diseases interfering with their metabolism e.g. untreated myxoedema, Cushing's syndrome, Type 1 diabetes mellitus, significant neurological or psychiatric illness such as epilepsy, schizophrenia, depression, eating disorders such as bulimia.
* Patients with Type 2 diabetes mellitus are ineligible unless anti-diabetic medication was not deemed necessary by the investigator and fasting (venous or arterialized capillary full blood from finger or ear) blood glucose > 6.1 mmol/l at screening. Re-test is allowed if first measure is above inclusion value. The corresponding exclusion criteria for plasma glucose is 7.0 mmol/l
* Patients currently (within the past 2 months) known to abuse or to be dependent on any drug, including alcohol (weekly consumption > 21 units of alcohol (men) or >14 units of alcohol (women))
* Hepatic or renal dysfunction (ASAT and/or ALAT > 2 x ULN and creatinine clearance < 30 mL/min estimated by central laboratory using Cockcroft and Gault formula, respectively)
* Known untreated hypercholesterolaemia (> 7 mmol/l). Patients with well regulated cholesterol using drugs for hypercholesterolaemia are allowed inclusion
* Known untreated hypertriglyceridaemia (> 3 mmol/l). Patients with well regulated triglyceride levels using drugs for hypertriglyceridaemia are allowed inclusion
* Drug treated thyroid diseases (well substituted hypothyroidism is allowed)
* Patients who suffer from hyperthyroid disease are not allowed in the study, even though they may be well treated by drugs
* Patients, who have recently diagnosed, not yet stable hypothyroid disease are not allowed in the study
* Patients who suffer from longstanding stable hypothyroid disease, well treated substitution are allowed to be included including hypothyroidism as a sequelae to definitive treatment of hyperthyroidism by surgery or radioactive iodine
* Malabsorptive intestinal disorders that can be assumed to affect the absorption of tesofensine
* Special diets (e.g., vegetarian, Atkins)
* Patients planning major changes in physical activity during the study to an extent that may interfere with the study outcome, as judged by the investigator
* Weight change of > 3 kg within 2 months prior to screening
* Mental or psychiatric disorder based on medical history only
* Surgically treated obesity
* Patients with systemic infections or inflammatory diseases
* History or presence of significant cardiovascular disease such as heart failure, ischemic heart disease, stroke, transient ischemic attacks
* Significant abnormalities on the ECG. according to the investigators opinion. Additional exclusionary ECG values: QTcB > 480 milliseconds (ms), PR interval > 240 ms, QRS interval > 120 ms
* Hypotension (i.e. supine systolic BP < 90 mm Hg) and/or symptomatic orthostatic hypotension (clinical symptoms of orthostatic hypotension associated with a decline ≥ 20 mm Hg in systolic BP at one minute after standing compared with the previous supine systolic BP obtained after 5 minutes of quiet rest) at screening visit
* Uncontrolled hypertension (i.e. sitting diastolic BP ≥ 95 mm Hg and sitting systolic BP ≥ 155 mm Hg) despite treatment for > 4 weeks prior to the screening visit as well as HR>90 bpm
* Known HIV infection (no tests required)
* Serologic evidence of active hepatitis B and/or C
* History of cancer within the past 5 years, excluding treated basal cell carcinoma
* Clinically significant or potentially disabling eye disorder, including uncontrolled glaucoma
* Current treatment with medication with known ocular toxicity such as chloroquine and hydroxychloroquine is prohibited
* Patients previously treated with tesofensine
* Patients treated with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Percent change and absolute change in body weight

SECONDARY OUTCOMES:
Waist circumference, waist-hip ratio, change in BMI, Sagittal diameter and DEXA
blood tests (Triglycerides, Cholesterol-total, LDL-C, HDL-C, LDH, Blood glucose fasting, HbA1c, C-reactive protein, Insulin and Adiponectin )
data from questionnaires (Baecke Questionnaire, Satiety & Appetite Questionnaire, POMS, and Impact of Weight on Quality of Life Questionnaire -Lite Version (IWQOL-Lite))
Safety & Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Arne V Astrup, MD, Principal Investigator — Department of Human Nutrition, The Royal Veterinary & Agricultural University
Locations (1):
- NeuroSearch A/S, Ballerup Municipality, Denmark

REFERENCES:
- [Background] Expression of concern--effect of tesofensine on bodyweight loss, body composition, and quality of life in obese patients: a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Apr 6;381(9873):1167. doi: 10.1016/S0140-6736(13)60778-3. No abstract available. PMID 23561987
- [Derived] Gilbert JA, Gasteyger C, Raben A, Meier DH, Astrup A, Sjodin A. The effect of tesofensine on appetite sensations. Obesity (Silver Spring). 2012 Mar;20(3):553-61. doi: 10.1038/oby.2011.197. Epub 2011 Jun 30. PMID 21720440
- [Derived] Astrup A, Madsbad S, Breum L, Jensen TJ, Kroustrup JP, Larsen TM. Effect of tesofensine on bodyweight loss, body composition, and quality of life in obese patients: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Nov 29;372(9653):1906-1913. doi: 10.1016/S0140-6736(08)61525-1. Epub 2008 Oct 22. PMID 18950853